CLINICAL TRIAL: NCT02745548
Title: Investigating Radiation-Induced Injury to Airways and Pulmonary Vasculature in Lung Stereotactic Ablative Body Radiotherapy (SAbR)
Brief Title: Bronchial Mapping (GCC 1635)
Status: Terminated | Type: Observational
Why Stopped: Grant ended, slow accrual- enrollment goal not met.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00069334
Record Dates: First submitted 2016-04-08; First posted 2016-04-20 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Cancer
Keywords: Lung Cancer; NSCLC (Non Small Cell Lung Cancer); SABR (Stereotactic ablative radiotherapy)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
In order to better understand radiation-induced lung toxicity, the investigator proposes a novel functional avoidance approach that incorporates central as well as peripheral BSS segments in the treatment planning process in order to quantify and account for their respective radiosensitivities. Specifically, the investigator proposes a systematic study that involves acquiring pre- and post-SAbR high-resolution CT and SPECT V/Q scans from lung cancer patients who receive radiotherapy, followed by auto-segmentation of the BSS elements using virtual bronchoscopy.

DETAILED DESCRIPTION:
Very few recent lung cancer therapies have had as positive an impact on public health as lung SAbR. Lung SAbR involves the precise administration of very high, biologically potent doses (54-70 Gy) in 3-5 fractions. The most recent update of the Radiation Therapy Oncology Group (RTOG) 0236 Phase II multi-center lung SAbR trial showed 5-year primary tumor control >90% in inoperable Stage I NSCLC patients with tumors ≤ 5cm. However, the use of such highly potent doses puts patients at risk for collateral toxicity including radiation pneumonitis and radiation injury to airways, causing stenosis, atelectasis and ultimately fibrosis. A review of 35 early-stage NSCLC SAbR clinical studies found that the reported maximum values of Grade ≥3 toxicities were between 10-28%. In the RTOG 0236 trial, 17% patients presented Grade ≥3 toxicities. Furthermore, toxicity has been shown to increase dramatically for centrally-located and/or larger (> 5cm) early-stage tumors. Due to these concerns, in current clinical practice, the use of high-dose-per-fraction lung SAbR is routinely indicated only for a small percentage (~3 - 4%) of the NSCLC population - inoperable, early-stage patients with small, peripheral lesions. Inoperable patients with early-stage central and/or larger tumors, higher stage and/or multiple lesions, and pulmonary oligometastases (metastatic disease that is limited in number of lesions and sites) are either treated with conventional radiotherapy and/or chemotherapy (~30 - 40% 5-year survival), or not treated (median survival ~1 year).

The segmented structures will be imported into a clinical radiotherapy treatment planning system in order to calculate dose to individual BSS elements. Follow-up CT images and follow-up SPECT V/Q scans will be used to characterize the radiosensitivity of these structures and spatially map the potential radiation-induced loss of lung function. Eventually, using this information, the investigator will investigate treatment planning strategies that help limit radiation dose and consequent damage to BSS elements, thereby reducing lung toxicity. The investigator hypothesizes that - Anatomically variable radiation injury to the bronchial tree and pulmonary vasculature is an important determinant of post-SAbR pulmonary toxicity and residual pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or metastatic lung lesions to be treated using stereotactic ablative radiotherapy (There is no limitation on the location or number of lesions for this study) OR Conventionally fractionated RT patients with primary or metastatic lung lesions
* Age ≥ 18 years. No gender or ethnic restrictions.
* Performance status ECOG ≥ 3
* Ability to hold breath for ~20 seconds
* Ability to understand and the willingness to sign a written informed consent.
* Any types and amounts of prior therapy will be allowed for this study.
* Maximum PTV dimension ≤ 70 mm

Exclusion Criteria:

* Children (age <18 years).
* Women who are pregnant, nursing, or trying to get pregnant.
* ECOG performance status < 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Thoracic malignancies who consent to recieving Radiation treatment at the University of Maryland, Baltimore, will be offered this protocol design.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Number of patients that show an association between radiation-induced collapse of branching serial structures elements and localized change in pulmonary function | 3 years
  Evaluating the association of RT and how branching structures change in lung function
Radiosensitivity of peripheral BSS segments in terms of dose dependent probability of collapse. | 3 years
  Evaluating the difference between dose and segmental collapse with pre- and post treatment MRI's

SECONDARY OUTCOMES:
Number of patients analyzed for creation of intensity modulated radiotherapy treatment plans that incorporate radiation dose thresholds for BSS elements | 3 years
  Evaluating IMRT plans incorporated radiation dose thresholds for BSS elements

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sawant, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No